CLINICAL TRIAL: NCT03090542
Title: 39 Day Randomized, Open Label, Two Arm Cross Over Study of Clinoptilolite (Gpur) in Healthy Adult Subjects Not Requiring or Receiving Lipid Lowering Therapy
Brief Title: GPur- Luminating Oral Cholesterol Kinetics Pilot Study
Acronym: GLOCK-pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Collaborative Research Network (Other)
Collaborators: GLOCK HEALTH, Science and Research, G.m.b.h. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GLOCK-Pilot 2017
Record Dates: First submitted 2017-03-06; First posted 2017-03-24 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Cholesterol Absorption
MeSH Terms: interventions — clinoptilolite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Product (Active Comparator)
  Interventions: Dietary Supplement: clinoptilolite

INTERVENTIONS:
Dietary Supplement: clinoptilolite — randomized, open-label, cross-over study of control vs clinoptilolite with a washout period separating the 2 phases
  Arms: Product

SUMMARY:
In healthy subjects not receiving or requiring lipid lowering therapy and who do not have diabetes, the use of clinoptilolite (GPUR) will result in a reduction of absorbed dietary cholesterol observed over 6 days of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age
* Not receiving or requiring lipid lowering therapy
* Willingness to give informed consent
* Able to keep a dietary log
* Willing to maintain a consistent day to day routine during the study (no major changes in lifestyle, exercise, food pattern, smoking habits, etc)

Exclusion Criteria:

* Current use of oral lipid binding agents (colesevelam, cholestyramine, ezetimibe) fibrates, niacin or statins
* Current use of dietary supplements enriched with fat soluble vitamins, mono/polyunsaturated fat (fish-oil etc.) or probiotics
* Any oral antibiotic use, currently or within the past 14 days
* Diabetes, Type I and Type II
* Currently following a restrictive diet
* GI motility disorders (irritable bowel syndrome, diabetic gastroparesis, etc)
* Prior gastric or bowel resection
* Inflammatory bowel disease (Crohns, ulcerative colitis, diverticulitis, celiac sprue, etc)
* Co-morbidities with anticipated life expectancy < 12 months
* ESRD on dialysis
* Known intolerance to silicium or aluminum compounds
* Excess alcohol consumption (>1 drink per day)
* Pregnancy, nursing or not taking/using contraception
* Hepatobiliary disorders or renal disease
* Plasma total cholesterol > 240mg/dl or Triglycerides > 265.5 mg/dl
* No plant-sterol enriched food products allowed in diet & supplements
* BMI > 35

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Percent change in fractional cholesterol absorption in human subjects taking clinoptilolite over 6 days | 39 days
  Primary Objective

SECONDARY OUTCOMES:
Percent change from baseline by gender to determine gender difference in fractional cholesterol absorption rates | 39 days
  Secondary Objective
Percent change from baseline to end of treatment to evaluate for safety changes in metabolic profile measurements | 39 days
  Secondary Objective

CONTACTS AND LOCATIONS:
Overall Officials: Narendra Singh, MD, Principal Investigator — Canadian Collaborative Research Network
Locations (1):
- Atlanta Heart Specialists, Cumming, Georgia, United States

IPD SHARING:
Plan to Share IPD: No